CLINICAL TRIAL: NCT01949571
Title: Phase II Clinical Studies on Anti-addictive Therapeutic Effects of Mirtazapine in Human Subjects Addicted to Cocaine.
Brief Title: Clinical Studies on the Therapeutic Effects of Mirtazapine on Drug-craving in Cocaine Addicts.
Acronym: MADC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Responsible Party: Principal Investigator, Dr Benito Antón Palma, Investigador en Ciencias Médicas "F"., Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: INPRF-01-MIR
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Drug-withdrawal.; Drug Abuse; Drug-induced Depressive State; AOD Craving; AODR Depressive State
Keywords: Mirtazapine.; Addiction.; Cocaine.; Cocaine-craving.; Cocaine-withdrawal
MeSH Terms: conditions — Substance Withdrawal Syndrome; Substance-Related Disorders; Behavior, Addictive | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mirtazapine (Experimental): During the first and second phase of the study, subjects assigned to the control group received one tablet of placebo under daily basis, whereas the mirtazapine group received 30 mg of mirtazapine daily. During the third phase, placebo group received same tablet under daily basis, whereas the mirtazapine group received 15 mg of mirtazapine.
  Interventions: Drug: Mirtazapine (REMERON, Schering-Plough-Organon)

INTERVENTIONS:
Drug: Mirtazapine (REMERON, Schering-Plough-Organon) — During the first and second phase of the study,the mirtazapine group received 30 mg of mirtazapine daily. During the third phase, the mirtazapine group received 15 mg of mirtazapine.
  Other Names: MIR

SUMMARY:
INTRODUCTION. One of the main problems of the treatment of cocaine-dependent patients is the high rate of relapses occurs within the first months after detoxification. In the early withdrawal phase, patients suffer severe anxious depressive symptoms, known in the argot as crash, which occurs in parallel with an appetite overflowed by re-experiencing the effects of the substance, known as craving. Most of the times, these clinical symptoms act as negative reinforcement, which can be severe enough to induce a drug-relapse that greatly hampers the treatment.

TYPE OF STUDY randomized, double-blind, placebo-experimental. GENERAL PURPOSE To determine the efficacy of mirtazapine for the treatment of cocaine dependence. SPECIFIC OBJECTIVES 1) To evaluate the efficacy in the treatment of craving in individuals with cocaine dependence disorder treated with mirtazapine during acute withdrawal phase. 2) Determine the efficacy of reducing anxious depressive symptomatology (Crash) associated with acute withdrawal in subjects with cocaine dependence disorder treated with mirtazapine. 3) Evaluate the maintenance of abstinence in patients with cocaine dependence disorder treated with mirtazapine. 4) Determine the efficacy of mirtazapine in the treatment of subjects dependent on cocaine comorbid with major depressive disorder.

HYPOTHESIS For pharmacokinetics and pharmacodynamics mirtazapine contribute to the reduction in the intensity of withdrawal symptoms in cocaine dependent subjects by acting on the neurochemical circuitry involved in the reward-seeking behavior and has a prolonged effect anticraving. METHOD The attending physician outpatient identifies the Addiction Clinic of the National Institute of Psychiatry who meet the inclusion criteria and invite them to participate voluntarily. If patients accept, send them to the principal investigator for the start of the ratings. Demographics INSTRUMENTS, MINI structured interview, Anxiety and Depression Scale Beck Scale.

DETAILED DESCRIPTION:
Evaluation. Evaluation of cocaine craving was assessed weekly through the Cocaine Craving Questionnaire (CCQ-G) (43-46). The CCQ-G measures the desire or urge level for drug consumption throughout the 45 Likert items established in the Questionnaire. The Likert scale consisted of seven options ranging from 1 to 7. Indicating from the lowest number (1) complete disagree of questions asked/item and the highest number (7) complete agreement of questions answered/item. CCQ-G items were written in past tense, with the intention that participants could report their cocaine craving status (level) during the previous week. Main items in the CCQ-G used to assess cocaine craving defined as factors were; a). Elements that denote intense cocaine craving (factor 1); b). Items that related to the anticipation of positive results (factor 2); c). Anticipation of relief from drug-withdrawal symptoms (factor 3); and d). Items that perceived a lack of control over cocaine consumption, denoting the intention and planning for cocaine consumption (factor 4).

Each week patient were assessed about their psychopathological status through the Symptom Check List 90 (SCL-90-R) (47-50). The SCL-90 evaluate the psychological degree of "distress" shown by a subject through 90 Likert-type reagents, ranging from 0 up to 4, and grouped into nine dimensions, which include, somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism.

Statistical Analysis.

Data were expressed, as mean ± SEM. To determinate the differences in score between groups over time, the data were then analyzed by a two-way repeated measures ANOVA with time (week) as the repeated measure. If there was a significant interaction between time and treatment, we then performed a Tukey's post-hoc test to detect significant differences between each one of the factors at each experimental phase. Comparisons between mean score obtained during each phase were analyzed by a two-way ANOVA (treatment x phase) followed by Tukey's test for post-hoc comparisons. The level of statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Who can read and write. Meet the DSM IV TR criteria for substance dependence disorder (Snuff, cocaine, ethanol and polysubstance.). That meet the ratings.

Exclusion Criteria:

disorder subjects with a history of dependency that are not abstinent (³. 1 month). Subjects with a history of neurological diseases. Subjects with general medical illness (eg CVD, hypertension, DM). Subjects prior to the implementation of neurocognitive testing report having consumed coffee, tea, alcohol or smoked three hours conducting assessments. Subjects who take more than 3 prescription drugs. Those who report being too tired. Subjects who report not having made an effort to answer the tests.

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2007-01; Primary Completion 2011-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Evidence that Mirtazapine attenuates cocaine-craving. | Four years

CONTACTS AND LOCATIONS:
Overall Officials: Benito Antón-Palma, MD-PhD, Study Director — National Institute of Psychiatry; Ricardo Nanni-Alvarado, Psychiatry, Principal Investigator — National Institute of Psychiatry
Locations (1):
- National Institute of Psychiatry, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Afshar M, Knapp CM, Sarid-Segal O, Devine E, Colaneri LS, Tozier L, Waters ME, Putnam MA, Ciraulo DA. The efficacy of mirtazapine in the treatment of cocaine dependence with comorbid depression. Am J Drug Alcohol Abuse. 2012 Mar;38(2):181-6. doi: 10.3109/00952990.2011.644002. Epub 2012 Jan 5. PMID 22221171
- [Background] Zueco Perez PL. [Mirtazapine in the treatment of cocaine-dependence in patients with methadone]. Actas Esp Psiquiatr. 2002 Nov-Dec;30(6):337-42. Spanish. PMID 12487943
- [Background] Graves SM, Rafeyan R, Watts J, Napier TC. Mirtazapine, and mirtazapine-like compounds as possible pharmacotherapy for substance abuse disorders: evidence from the bench and the bedside. Pharmacol Ther. 2012 Dec;136(3):343-53. doi: 10.1016/j.pharmthera.2012.08.013. Epub 2012 Aug 29. PMID 22960395